CLINICAL TRIAL: NCT05197036
Title: A Multi-Centre Study in Patients Undergoing Total Knee Replacement With Smith+Nephew Porous Total Knee Arthroplasty (TKA) System
Brief Title: A Global Clinical Study Investigating the Safety and Effectiveness of Smith and Nephew's Porous Knee System in Patients Who Need a Total Knee Replacement Due to Degenerative Arthritis, Post-traumatic Arthritis or Inflammatory Arthritis
Status: Active, not recruiting | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: POROUS.TKA.SYSTEM.2021.07
Record Dates: First submitted 2022-01-04; First posted 2022-01-19 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Osteoarthritis; Post-traumatic Arthritis; Rheumatoid Arthritis
Keywords: Arthritis; Osteoarthritis; Rheumatoid Arthritis; Post-traumatic Arthritis; Total Knee Arthroplasty (TKA); Knee Replacement; Cementless; Knee; Smith and Nephew
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Arthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LEGION Porous CR with Hydroxyapatite: Patients who have already received or a due to receive a Porous Tibia + LEGION Porous CR with HA femoral component (min 117 subjects)
  Interventions: Procedure: Total Knee Arthroplasty
- LEGION Porous CR without Hydroxyapatite: Patients who have already received or a due to receive a Porous Tibia + LEGION Porous CR without HA femoral component (min 117 subjects)
  Interventions: Procedure: Total Knee Arthroplasty

INTERVENTIONS:
Procedure: Total Knee Arthroplasty — A surgical procedure to replace both the tibial and femoral articular surfaces with titanium prostheses.
  Other Names: Total Knee Replacement

SUMMARY:
A clinical trial investigating the safety and effectiveness of Smith and Nephew's FDA-approved Porous Total Knee System, which is used to replace worn away and diseased knee joints. The aim of this study is to show that most patients who receive the Porous Total Knee System have reduced pain, greater mobility and a long-lasting implant post-surgery.

DETAILED DESCRIPTION:
Patients who need a total knee replacement or have recently had a total knee replacement with the Smith and Nephew Porous Total Knee System will be enrolled into the study. Before surgery X-rays will be collected and questionnaires will be administered which ask the patient about knee pain, activities of daily living, quality of life and how they feel about their knee. The same X-rays and questionnaires will be asked before surgery and then after surgery at various intervals up to 10 years post-surgery.

ELIGIBILITY:
Inclusion Criteria:

1. A) Subject needing primary TKA due to degenerative joint disease (primary diagnosis of osteoarthritis), post-traumatic arthritis or inflammatory arthritis.

   OR

   B) Subject has undergone primary TKA with Smith+Nephew Porous knee system in past 12 months to repair degenerative joint disease, post- traumatic arthritis or inflammatory arthritis and all the following conditions have been met:
   * Preoperative KOOS JR and radiographs have been obtained
   * 6-Month KOOS JR and radiographs have been obtained or these can be collected prospectively in window per schedule of events
2. Subject agrees to consent and to follow the prospective study visit schedule (as defined in the study protocol and informed consent form) by signing the Independent Review Board (IRB)/Independent Ethics Committee (IEC) approved informed consent form.
3. Subject is willing to attend study follow-up visits for up to five (5) years post-surgery.
4. Subject is able to read, understand, and communicate responses to Patient Reported Outcome assessments.
5. Subject is 18-80 years old (inclusive).

Exclusion Criteria:

1. Subject received TKA on the contralateral knee as a revision for a previously failed total or unicondylar knee arthroplasty.
2. Subject has a Body Mass Index (BMI) ≥ 40 at time of surgery.
3. Subject has ipsilateral hip arthritis resulting in flexion contracture.
4. At the time of enrolment, subject has one or more of the following arthroplasties that are not fully healed and well-functioning, as determined by the investigator: Ipsilateral or contralateral primary total hip arthroplasty or hip resurfacing arthroplasty; Contralateral primary total knee or unicondylar knee arthroplasty.
5. Subject has a condition that may interfere with the TKA survival or outcome (e.g. Paget's or Charcot's disease, vascular insufficiency, lupus, muscular atrophy, uncontrolled diabetes, moderate to severe renal insufficiency or neuromuscular disease).
6. Subject has a known allergy to one or more of its components of the study device.
7. Any subject with hardware present in distal femur or proximal tibia.
8. Any subject that meets the definition of a Vulnerable Subject per ISO 14155 Section 3.55.
9. Subject is entered in another drug, biologic, or device study or has been treated with an investigational product in the past 30 days.
10. Subject, in the opinion of the Investigator, has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study including mental illness, drug or alcohol abuse.
11. Subject is known to be at risk for lost to follow-up, or failure to return for scheduled visits.
12. Women who are pregnant, nursing, or of child-bearing potential who are not utilizing highly effective birth control measures.
13. Subjects who have participated previously in this clinical trial and who have been withdrawn.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient population will be selected by investigators from their clinics. Patients who report pain/mobility issues and who have been recommended for total knee replacement with Porous Total Knee System by their surgeon.
Sampling Method: Non-Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2026-06-19 (Estimated); Study Completion 2033-12-25 (Estimated)

PRIMARY OUTCOMES:
Implant Survivorship (femoral and/or tibial component) 2 Years Post-Surgery | 2 years post-surgery
  Survivorship of the femoral and/or tibial component of the implant is defined as the cumulative proportion of femoral and/or tibial components without a revision.

SECONDARY OUTCOMES:
Patient Reported Outcomes - Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS JR) | Pre-op, 6 weeks, 6 months, 2 years, 3 years, 5 years and 10 years
  KOOS JR assesses patient stiffness (1 item), pain (4 items), and functions of daily living (2 items). Scores range from 0 to 100 with a score of 0 indicating total knee disability and 100 indicating perfect knee health.
Patient Reported Outcomes - Oxford Knee Score (OKS) | Pre-op, 6 weeks, 6 months, 2 years, 3 years, 5 years and 10 years
  The OKS contains 12 equally weighted questions on activities of daily living. Responses to each question range from 0-4 with a range of a possible overall score from 0-48. A score of 0 is the worst possible outcome while a score of 48 is the best possible outcome.
Patient Reported Outcomes - Forgotten Joint Score (FJS) | Pre-op, 6 weeks, 6 months, 2 years, 3 years, 5 years and 10 years
  The FJS questionnaire focuses on the study participant's awareness of a specific joint in everyday life. Joint awareness can be simply defined as any unintended perception of a joint. The FJS for an individual participant is rated on a scale of 1-100 where 100 is the best/max score.
Radiographic Assessment - Implant Position | 6 months, 2 years, 5 years and 10 years
  Implant position will be assessed by the femoral flexion angle, tibial angle, and posterior tibial slope angle from AP and lateral radiographs.
Radiographic Assessment - Implant Migration | 6 months, 2 years, 5 years and 10 years
  Migration will be assessed in accordance with the following definitions:
  * 0. Absent: Absence of progressive radiolucency OR absence of movement of the implant.
  * 1. Present: Presence of progressive radiolucency AND presence of movement of the implant.
Radiographic Assessment - Progressive Radiolucency | 6 months, 2 years, 5 years and 10 years
  Progressive Radiolucency will be assessed in accordance with the following definitions:
  * 0. Absent: No evidence of progressive radiolucency at the bone-cement interface relative to the last measured Radiolucent Line time point.
  * 1. Present: Presence of an increase >1 mm of the Radiolucent Line (Bone-Cement) width and/or new involvement of additional component zones relative to the last measured Radiolucent Line time point.
Radiographic Assessment - Implant Loosening | 6 months, 2 years, 5 years and 10 years
  Both aseptic and septic component loosening will be evaluated to assess loss of implant fixation with the following definitions:
  * 0. Absent: No evidence of specific imaging features of loosening in the joint space.
  * 1. Present: Presence of apparent imaging features of loosening in the joint space.
Post-Operation Device Related Re-Interventions Related to Operative Knee | Post-op through study completion, approximately 10 years
  Count of device-related re-interventions that occur related to the operative knee post-operation.
Implant Survival Rate Up to 10 Years Post-Operation | 1 year, 2 years, 5 years and 10 years
  Survivorship of the implant will be defined as the cumulative proportion of all knee implant components without a revision.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Kamali, Study Director — Smith & Nephew, Inc.
Locations (18):
- United States (12):
  - Emory Orthopaedics and Spine Hospital, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Core Institute, Novi, Michigan
  - Syracuse Orthopedic Specialists, East Syracuse, New York
  - NYU Langone Health Orthopedic Hospital, New York, New York
  - Columbia University, New York, New York
  - Duke Health, Morrisville, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Erlanger Health, Chattanooga, Tennessee
  - UTHealth, Houston, Texas
  - University of Wisconsin, Madison, Wisconsin
- Australia (2):
  - St George and Sutherland Centre for Clinical Orthopaedic Research, Sydney, New South Wales
  - The Avenue Hospital, Windsor, Victoria
- Concordia Joint Replacement Group, Winnipeg, Manitoba, Canada
- Netherlands (2):
  - Medical Center Leeuwarden, Leeuwarden, Leeuwarden
  - Sint Maartenskliniek, Ubbergen, Ubbergen,
- Umeå University Hospital, Umeå, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Undecided